CLINICAL TRIAL: NCT05442918
Title: Expected Normal Ketone Values After Very Low and Bariatric Surgery
Status: Completed | Type: Observational
Sponsor: St Vincent's Hospital Melbourne (Other)
Responsible Party: Principal Investigator, Michael Hii, Doctor, St Vincent's Hospital Melbourne
Other Study IDs: StVincentsMelbourne
Record Dates: First submitted 2022-06-26; First posted 2022-07-05 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Diabetes Mellitus; Ketoacidosis
MeSH Terms: conditions — Diabetes Mellitus; Ketosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- General Surgery: All patients undergoing either elective laparoscopic/open cholecystectomy, laparoscopic/open hiatus hernia repair, laparoscopic/open inguinal hernia repair, laparoscopic/open umbilical hernia repair or laparoscopic ventral wall hernia repair.
- Bariatric Surgery: Participants undergoing elective bariatric surgery (laparoscopic sleeve gastrectomy or roux-en-y gastric bypass). Those in the bariatric arm must have been on a VLCD pre operatively

SUMMARY:
The investigators propose a multicenter prospective study in patients undergoing either an elective bariatric procedure or an elective benign procedure, including laparoscopic/open cholecystectomy, laparoscopic/open hiatus hernia repair, laparoscopic/open inguinal hernia repair, laparoscopic/open umbilical hernia repair or laparoscopic ventral wall hernia repair. Perioperative blood ketone and venous blood gas levels will be measured pre-surgery, post-surgery and on post-operative days until discharge.

Our primary research objective is to clarify the expected perioperative ketone and blood gas levels in elective bariatric patients who have been on a VLCD and fasting for surgery, compared to elective surgical patients who have only been fasting prior to surgery.

DETAILED DESCRIPTION:
Bariatric surgery is fast becoming a mainstream option for achieving long-term weight loss in the morbidly obese population due to the paucity of other effective alternatives. It is indicated in those with a Body Mass Index (BMI) >40, or those with an obesity-related comorbidity with a BMI >35. One of the most common of these comorbidities is Type 2 Diabetes Mellitus (T2DM).

In the weeks preceding bariatric surgery, it is routine for patients to be placed on a very low calorie diet (VLCD). The aim is to reduce abdominal wall thickness, visceral adiposity and hepatomegaly. Overall, this contributes to reduced technical difficulties at operation.

VLCD achieve rapid weight loss in the short term by inducing ketosis. This is achieved by reducing the consumption of carbohydrate and fat, while increasing protein intake. The depletion of caloric intake leads to decreased glucose stores. This then leads to a metabolic shift towards production of ketone bodies, which are produced by the liver via the oxidation of fatty acids. Ketones are then transported to tissue to take over the role of glucose as the main energy source for the central nervous system. The objective is to reduce fat mass without causing excess loss of muscle mass.

Overall the VLCD regime, via the induction of ketosis, is very successful in weight reduction. However this mechanism of action, and the production of ketone bodies, is now being questioned in those prescribed a new class of glucose lowering medication used to treat T2DM.

Sodium-glucose co-transporter-2 (SGLT2) inhibitors, also called gliflozins, are medications that reduce absorption of glucose in the kidney thus increasing excretion via urine. Phase 3 trials have shown them to be safe for treatment of T2DM however; however concern has been raised about development of a euglycaemic diabetic ketoacidosis. It is thought to occur when stress hormones lead to increased ketosis in patients taking SGLT2 inhibitors, which appear to alter insulin production. This situation can occur in the perioperative period if the SGLT2 inhibitors have not been correctly withheld pre-operatively.

Current guidelines from the Australian and New Zealand College of Anaesthetists recommend the cessation of SLGT2 inhibitors 3 days prior to surgery. If this has not occurred, they state blood ketones should be tested. If the blood ketones are >0.6, it is a strong recommendation to postpone non-urgent surgery. Ketone and base excess levels are then used to monitor patients in the perioperative period.

The confounding factor in these patients now presents itself- what are the expected blood ketone levels in bariatric patients who have been on two week of pre-operative VLCD and are fasting for surgery?

ELIGIBILITY:
Inclusion Criteria:

General surgery group, undergoing the following elective surgeries:

* laparoscopic/open cholecystectomy
* laparoscopic/open hiatus hernia repair
* laparoscopic/open inguinal hernia repair
* laparoscopic/open umbilical hernia repair
* laparoscopic ventral wall hernia repair

Bariatric surgery group, undergoing the following elective surgeries and a very low calorie diet before surgery:

* laparoscopic sleeve gastrectomy
* laparoscopic roux-en-y gastric bypass

Exclusion Criteria:

* currently on SLGT2 inhibitor
* non English speaking
* procedure abandoned

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients undergoing either elective laparoscopic/open cholecystectomy, laparoscopic/open hiatus hernia repair, laparoscopic/open inguinal hernia repair, laparoscopic/open umbilical hernia repair or laparoscopic ventral wall hernia repair or elective bariatric procedure will be recruited consecutively. Those in the bariatric arm must have been on a VLCD pre operatively. Recruitment does not require blinding or randomization.
  Patients will be excluded if they are non-English speaking or cannot consent to the project, if they are already taking an SLGT2 inhibitor or if their procedure was abandoned.
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-12-11 (Actual); Study Completion 2020-12-12 (Actual)

PRIMARY OUTCOMES:
Blood ketone | Immediately prior to surgery, immediately post-surgery, daily until discharge until up to 1 week
  blood ketone levels
Venous blood gas levels | Immediately prior to surgery, immediately post-surgery, daily until discharge until up to 1 week
  Primary outcome measures are blood ketone, and venous blood gas levels.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hii, FRACS, Principal Investigator — St Vincent's Hospital Melbourne
Locations (1):
- St Vincent's Hospital Melbourne, Fitzroy, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Mollah T, Gillespie C, Cocco A, Taylor L, Chong L, Hii MW. Defining Physiological Ketosis Following Very-Low-Calorie Diets. J Surg Res. 2023 Oct;290:197-202. doi: 10.1016/j.jss.2023.05.001. Epub 2023 Jun 2. PMID 37271067